CLINICAL TRIAL: NCT06817369
Title: The Effect of the Training Given by Using Internal and External Focus on the Sportive Performance of Girl Volleyball Players
Brief Title: Internal or External Focus in Girl Volleyball Players?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gizem Gul Turan, PhD student and Lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Girl Volleyball Player
Record Dates: First submitted 2024-01-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-01

CONDITIONS: Internal and External Focus
Keywords: internal focus; external focus; volleyball players; sport; motor learning

STUDY DESIGN:
Intervention Model Description: A two-arm parallel task involves two groups of participants. While the first group receives exercise training with an internal focus, the other group receives exercise training with an external focus. Therefore, during the experiment, the participants in the first group receive exercise training with internal focus "in parallel" with the participants in the other group who receive exercise training with external focus.Randomization will be done randomly.
Who Masked: Investigator
Masking Description: Participants in two groups randomly allocated by the researcher will not know which group they belong to, but the researcher will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Internal focus) (Experimental): Jump evaluation will be made using the Vertical Jump Test. Flamingo balance test will be used in static balance evaluation, and y balance test will be used in dynamic balance evaluation. Standard Sit-Reach Test will be used to evaluate the flexibility of the back and legs. Wall Catch Coordination Test will be used to evaluate hand eye coordination. Evaluations will be made before and after exercise There will be 5 exercises.
  Internal focus instructions will be applied while performing the exercises.
  Interventions: Other: Exercises given with internal focus instructions
- Group 2 (external focus) (Experimental): Jump evaluation will be made using the Vertical Jump Test. Flamingo balance test will be used in static balance evaluation, and y balance test will be used in dynamic balance evaluation. Standard Sit-Reach Test will be used to evaluate the flexibility of the back and legs. Wall Catch Coordination Test will be used to evaluate hand eye coordination. Evaluations will be made before and after exercise There will be 5 exercises. External focus instructions will be applied while performing the exercises
  Interventions: Other: Exercises given with external focus instructions

INTERVENTIONS:
Other: Exercises given with internal focus instructions — Both groups of girl volleyball players will be given 5 exercises. Exercise 1: Hands-free vertical jump (the movement of an individual jumping from a certain point and then jumping back to the same point) Exercise 2: Training in catching and throwing the ball thrown by the physiotherapist while the individual remains stationary for 30 seconds in the lunge position Exercise 3: Weight transfer on balance beam Exercise 4: Stretching the hamstring and trunk muscles / Bending the trunk while standing upright and touching the toes to the ground exercise Exercise 5: Exercise used in Wall Catch Coordination test Each exercise will be 3 sets of 10 repetitions / 1-2 minutes of rest between each set.
  Arms: Group 1 (Internal focus)
Other: Exercises given with external focus instructions — Both groups of girl volleyball players will be given 5 exercises. Exercise 1: Hands-free vertical jump (the movement of an individual jumping from a certain point and then jumping back to the same point) Exercise 2: Training in catching and throwing the ball thrown by the physiotherapist while the individual remains stationary for 30 seconds in the lunge position Exercise 3: Weight transfer on balance beam Exercise 4: Stretching the hamstring and trunk muscles / Bending the trunk while standing upright and touching the toes to the ground exercise Exercise 5: Exercise used in Wall Catch Coordination test Each exercise will be 3 sets of 10 repetitions / 1-2 minutes of rest between each set.
  Arms: Group 2 (external focus)

SUMMARY:
The subject of the research is to examine the effects of training given with internal and external focus on sports performance in young and adolescent girl volleyball players. The aim of this study is to compare the effects of training given with internal and external focus on balance, jumping, hand-eye coordination and flexibility in order to improve sports performance in young and adolescent girl volleyball players.Data will be collected between 01.02.2024-01.01.2025 from individuals who accepted the research in the junior and adolescent girls' volleyball team affiliated with the Malatya Provincial Directorate of the Ministry of Youth and Sports. The individuals in the junior and adolescent girls' volleyball team included in the study by the researchers will be randomly divided into 2 groups.A minimum of 15 people for each 2 groups will be included in the study. Balance, jumping, hand-eye coordination and flexibility training using internal focus for the 1st group. The second group will be given balance, jumping, hand-eye coordination and flexibility training using external focus. In the study, both groups will receive the same exercise training, for the same duration and frequency. Only exercise management guidelines will be differentiated. Balance (static and dynamic), jumping performance, hand-eye coordination and flexibility will be evaluated before and after exercise training.

DETAILED DESCRIPTION:
Sports are activities that improve people's mental and physical characteristics and have multifaceted effects throughout life. These parts should be present in your life from an early age. Volleyball, with influences from different cultures and environments, especially from Turkey's most successful team sports, where women reach large masses. Volleyball is a dynamic team sport that involves very intense movements such as speed, jumping and changing direction. In volleyball, many motor skills need to be coordinated and trained effectively and developed. Basic motor skills in volleyball; Strength, endurance, endurance, coordination, speed and balance are maintained. Neurodevelopmental movement training given to the athlete according to motor learning geometry maximizes the athlete's sporting success and also positively affects their physical, mental and social development.

Motor learning is the process by which an individual develops motor skills and performs with a permanent change in performance that is acquired as a function of practice or experience. Instructions and complementary feedback are important influencing factors to support motor learning processes. Storing (re)motoring will be learned immediately, in case of registration, the accepted information will receive instructions on the correct movement system. These instructions typically refer to coordinating body movements, including the order, form, and timing of various limb movements. Instructions that direct the patient's attention to his own movements create an internal focus of attention. A simple change in the wording of instructions can have a significant impact on performance and learning. Transferring the patient's attention to the effects of his movements on the environment (external focus) is achieved through more effective and efficient movements.

There are studies in the literature comparing the frequency of internal focus and external focus when training sport-specific motor skills. In a distribution made, child athletes in internal and externally focused feedback groups performed free throw training, and a significant learning advantage was stated in the test results, considering the child athletes receiving externally focused feedback. Another reported that regular externally focused feedback did not increase the accuracy of the table tennis backhand stroke compared to internally focused feedback. In the literature, externally focused feedback was not found in local child athletes and novice athletes, where running was beneficial. Another study in the literature is external feedback in competitive girls' football volleyball players, and according to internal feedback, it is bet that the dunk speed in volleyball has an immediate performance on the athletes.

In general, studies in the literature have examined the effects of internal and external tension on volleyball-specific motor performance such as dunk speed and permanence vertical jump performance in girls' volleyball teams on the regime in certain age groups, but no comparison was found between groups. The investigators did not perform these operations but designed them based on the deficiencies in the literature.

The research was planned as an experimental study. The study will be carried out in two private sports clubs operating in Malatya, in the little girls' volleyball team between the ages of 7-11 and the adolescent girls' volleyball team between the ages of 12-14. The necessary permission to carry out the study will be obtained from the Malatya Provincial Directorate of the Ministry of Youth and Sports. The study will be carried out in accordance with the principles of the Declaration of Helsinki. By participating in the study, the parents/guardians of the children in the girls' volleyball team will be informed in detail about the study and their written consent will be obtained. Participating children's age, height, weight, age of starting sports, duration of participation in sports (month/day), frequency of participation in sports (day/week) will be questioned with the case report form.

Research Sample size: Type I error 0.05 on G-Power 3.1.7 package program (Heinrich-Heine-Universitat, Dusseldorf, Germany); Type II error was calculated by taking 0.2. The power of the test was determined as 0.8. In the study conducted, the minimum number of subjects required to be included in each group was calculated as 15 in order for the difference of 2.3 units regarding total game performance to be found significant.

Collection of Data Data will be collected between 01.02.2024-01.01.2025 from individuals who accepted the research in the junior and adolescent girls' volleyball team affiliated with the Malatya Provincial Directorate of the Ministry of Youth and Sports. The individuals in the junior and adolescent girls' volleyball team included in the study by the researchers will be randomly divided into 2 groups. Balance, jumping, hand-eye coordination and flexibility training using internal focus for the 1st group. The second group will be given balance, jumping, hand-eye coordination and flexibility training using external focus. In the study, both groups will receive the same exercise training, for the same duration and frequency. Only exercise management guidelines will be differentiated. Balance (static and dynamic), jumping performance, hand-eye coordination and flexibility will be evaluated before and after exercise training.

Reviews The equipment to be used for evaluations will be covered by the researcher. Participating children's age, height, weight, age of starting sports, duration of participation in sports (month/day), frequency of participation in sports (day/week) will be questioned with the case report form. Height will be measured with a stadiometer and weight with a 0.5 kg precision scale.

Jump evaluation will be made using the Vertical Jump Test. It is a test with a very high reliability coefficient (rxy=0.97) for determining the athlete's jumping force. The athlete reaches the maximum point he can reach with one arm in front of the platform to be tested and the distance is determined. The difference between this point where the athlete can reach and the highest point he can reach by jumping is determined and the height is recorded in cm. The test must be repeated twice to determine the best score.

Flamingo balance test will be used in static balance evaluation, and y balance test will be used in dynamic balance evaluation. Flamingo balance test is used to measure static balance. For this test, a balance board made in standard sizes determined by Eurofit is used. The balance board is made by mounting two wooden beams, 2 cm wide and 15 cm long, spaced apart and perpendicularly, under two wooden beams that are 4 cm thick, 3 cm wide and 30 cm long. The participants' ability to stand on one leg on the balance board is tested. The participant steps on the balance board with one foot and bends the knee while holding the free foot with the hand on the same side. Meanwhile, his free hand is supported by the tester. As soon as the participant feels that he has regained his balance, he releases the tester's hand and the stopwatch is started at that moment. If the held foot is released or if the balance is disturbed and the foot leaves the balance board, the stopwatch is stopped and the time is recorded. If the person being tested does not lose balance for 60 seconds, the test is terminated. Y balance test is a dynamic test performed in the standing position on one leg. It examines how the core area and both extremities work under body weight. Before the test, individuals remove their shoes and stand on the foot plate in the center of the Y Balance Test area. Individuals are then instructed to maintain a single-leg stance while reaching as far as possible with the opposite leg and return to the starting position on the middle 22 platform without losing balance. In the test, individuals are asked to reach the maximum distance in 3 directions (anterior, posteromedial and posterolateral), allowing 3 attempts for each leg. The maximum reach distance is recorded for each consecutive attempt.

The Standard Sit-Reach Test will be used to evaluate the flexibility of the back and leg. The child is seated on the ground on a flat surface, allowed to rest the soles of his bare feet flat on the test stand, then his body is extended forward as far as he can reach, and he is asked to wait for a second or two at the last point with the arms and fingers tense and straight, and after two attempts, he It is recorded well.

Wall Catch Coordination Test will be used to evaluate hand eye coordination. The participant stands facing the wall at a distance of 3 meters. The ball is thrown from bottom to top by keeping the shoulder stable, provided that it is caught with the throwing hand. After a certain number of trials, the other hand is tested. Scoring of successful shots is done the same way for both hands. To assist in evaluating the results, the score of the participant's preferred side should be recorded. A tennis or baseball ball can be used to perform the test.

treatments Exercises Exercise 1: Hands-free vertical jump (the movement of an individual jumping from a certain point and then jumping back to the same point) 3 sets of 10 repetitions / 1-2 minutes of rest between each set Internal Focus Instructions: With participants hands free, jump to the highest point participants can without disturbing participants body balance.

External Focus Instructions: With participants hands free, try to jump and touch the fixed bar.

Exercise 2: Training in catching and throwing the ball thrown by the physiotherapist while the individual remains stationary for 30 seconds in the lunge position / 3 sets of 10 repetitions / 1-2 minutes of rest between each set Internal Focus Instructions: While standing in the lunge position, hold the ball thrown by the physiotherapist without disturbing participants body balance and throw it back.

External Focus Instructions: While standing in the lunge position, catch the ball thrown by the Physiotherapist and throw it into the circle on the wall.

Exercise 3: Weight transfer on balance beam - 3 sets of 10 repetitions / 1-2 minutes rest between each set Internal Focus Instructions: Equalize the position of participants feet on the balance beam External Focus Instructions: Transfer the tilt of the bosun from right to left / left to right Exercise 4: Stretching the hamstring and trunk muscles / Bending the trunk while standing upright and touching the toes to the ground exercise - 3 sets of 10 repetitions / 1-2 minutes rest between each set Internal Focus Instructions: Bend participants torso, extend participants fingertips as much as possible, and feel the muscles on the back of participants legs tighten.

External Focus Instructions: Bend participants body and touch participants fingertips to the line on the floor.

Exercise 5: Exercise used in Wall Catch Coordination test / 3 sets of 10 repetitions / 1-2 minutes rest between each set Internal Focus Instructions: Throw the tennis ball against the wall in front of participants with one hand and try to catch it again with participants feet fixed on the ground without disturbing participants body balance.

External Focus Instructions: Try to hit the tennis ball with one hand into the ring on the wall in front of participants and hold it with the same hand.

ELIGIBILITY:
Inclusion Criteria:

* Being a volleyball player in the little/adolescent girls' volleyball team
* Having been participating in volleyball regularly for at least 6 months

Exclusion Criteria:

* Participating in more than one sport
* Having an orthopedic or neurological musculoskeletal disorder
* Having had a surgical operation within the last year

Ages: 7 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Girls will be included in the study.
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Effect of Different Focus Training (internal or external) on Jumping Performance in Girl Volleyball Players with Vertikal Jump Test | 1 week
  Jumping performance was evaluated using the Vertical Jump Test, with jump height recorded in centimeters; higher jumps indicated better performance. Measurements were taken before and after exercise training, and results were analyzed for each test separately.
Evaluation of the Effect of Different Focus Training (internal or external) on Statik Balance in Girl Volleyball Players with Flamingo Balance Test | 1 week
  Static balance was measured by the Flamingo Balance Test, with balance time in seconds; longer times reflected better balance. Measurements were taken before and after exercise training, and results were analyzed for each test separately.
Evaluation of the Effect of Different Focus Training (internal or external) on Dynamic Balance in Girl Volleyball Players with Y Balance Test | 1 week
  Dynamic balance was assessed using the Y Balance Test, with reach distances in three directions; longer distances indicated better balance. Measurements were taken before and after exercise training, and results were analyzed for each test separately.
Evaluation of the Effect of Different Focus Training (internal or external) on Flexibility in Girl Volleyball Players with Sit and Reach Test | 1 week
  Flexibility of the back and legs was tested with the Sit and Reach Test, recording forward reach in centimeters; greater distances reflected increased flexibility. Measurements were taken before and after exercise training, and results were analyzed for each test separately.
Evaluation of the Effect of Different Focus Training (internal or external) on Hand-eye coordination in Girl Volleyball Players with Wall Catch Coordination Test | 1 week
  Hand-eye coordination was evaluated by the Wall Catch Coordination Test, where more catches indicated better coordination. Measurements were taken before and after exercise training, and results were analyzed for each test separately.

SECONDARY OUTCOMES:
Evaluation of the effect of free vertical jump exercise training on jumping performance in girls volleyball players. | 1 week
  The girl volleyball players performed 5 different exercises. One of these was the free vertical jump exercise. The exercise was performed in 3 sets of 10 repetitions with 1-2 minutes of rest between sets. The exercise was performed with internal or external focus instructions and the effects of these instructions on the jumping performance of young girl volleyball players were examined. Which focus instruction was more effective will be determined by comparing the units (e.g. centimeters) of the vertical jump test measured before and after the exercise. The test will be compared with its own before and after values; the measurements will not be combined.
Evaluation of the effect of catching and throwing the ball in free lunge position on static balance in girl volleyball players | 1 week
  The girl volleyball players performed 5 different exercises. One of them was a lunge position, catching and throwing the ball. The exercise was performed in 3 sets of 10 repetitions, with 1-2 minutes of rest between sets. The exercise was performed with internal or external focus instructions, and the effects of these instructions on the static balance of young girl volleyball players were examined. Which focus instruction was more effective will be determined by comparing the flamingo balance test units (e.g. seconds) measured before and after the exercise. The test will be compared with its own before and after values; the measurements will not be combined.
Evaluation of the effect of weight transfer exercise on the bos on dynamic balance in girl volleyball players | 1 week
  Girl volleyball players performed 5 different exercises. One of them was a weight transfer exercise on the bos. The exercise was performed in 3 sets of 10 repetitions with 1-2 minutes of rest between sets. The exercise was performed with internal or external focus instructions and the effects of these instructions on dynamic balance of girl volleyball players were examined. Which focus instruction was more effective will be determined by comparing the Y balance test units (e.g. centimeters) measured before and after the exercise. The test will be compared with its own before and after values; the measurements will not be combined.
Evaluation of the effects of body bending and toe touching exercise on flexibility in girl volleyball players | 1 week
  The girls volleyball players performed 5 different exercises. One of them was the body bending and the finger touching the ground exercise. The exercise was performed in 3 sets of 10 repetitions and 1-2 minutes of rest was given between sets. The exercise was performed with internal or external focus instructions and the effects of these instructions on the flexibility of the girls volleyball players were examined. Which focus instruction was more effective will be determined by comparing the sit-and-reach test units (e.g. centimeters) measured before and after the exercise. The test will be compared with its own before and after values; the measurements will not be combined.
Evaluation of the effect of throwing the ball to the wall and catching it back exercise on hand-eye coordination in girl volleyball players | 1 week
  The girls volleyball players performed 5 different exercises. One of them was throwing the ball against the wall and catching it back. The exercise was performed in 3 sets of 10 repetitions, with 1-2 minutes of rest between sets. The exercise was performed with internal or external focus instructions, and the effects of these instructions on the hand-eye coordination of the girls volleyball players were examined. Which focus instruction was more effective will be determined by comparing the wall-catch coordination test units (e.g. catch count) measured before and after the exercise. The test will be compared with its own before and after values; the measurements will not be combined.

CONTACTS AND LOCATIONS:
Locations (1):
- Inönü University, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Wong TKK, Ma AWW, Liu KPY, Chung LMY, Bae YH, Fong SSM, Ganesan B, Wang HK. Balance control, agility, eye-hand coordination, and sport performance of amateur badminton players: A cross-sectional study. Medicine (Baltimore). 2019 Jan;98(2):e14134. doi: 10.1097/MD.0000000000014134. PMID 30633230
- [Background] Welling W, Benjaminse A, Gokeler A, Otten B. Enhanced retention of drop vertical jump landing technique: A randomized controlled trial. Hum Mov Sci. 2016 Feb;45:84-95. doi: 10.1016/j.humov.2015.11.008. Epub 2015 Nov 23. PMID 26615475
- [Background] Slovak L, Sarvestan J, Iwatsuki T, Zahradnik D, Land WM, Abdollahipour R. External focus of attention enhances arm velocities during volleyball spike in young female players. Front Psychol. 2023 Jan 5;13:1041871. doi: 10.3389/fpsyg.2022.1041871. eCollection 2022. PMID 36687905
- [Background] Niznikowski T, Luba-Arnista W, Arnista P, Porter JM, Makaruk H, Sadowski J, Mastalerz A, Niznikowska E, Shaw A. An external focus of attention enhances table tennis backhand stroke accuracy in low-skilled players. PLoS One. 2022 Dec 1;17(12):e0274717. doi: 10.1371/journal.pone.0274717. eCollection 2022. PMID 36455038
- [Background] Perreault ME, French KE. External-Focus Feedback Benefits Free-Throw Learning in Children. Res Q Exerc Sport. 2015;86(4):422-7. doi: 10.1080/02701367.2015.1051613. Epub 2015 Jul 31. PMID 26230869
- [Background] Gokeler A, Neuhaus D, Benjaminse A, Grooms DR, Baumeister J. Principles of Motor Learning to Support Neuroplasticity After ACL Injury: Implications for Optimizing Performance and Reducing Risk of Second ACL Injury. Sports Med. 2019 Jun;49(6):853-865. doi: 10.1007/s40279-019-01058-0. PMID 30719683
- [Background] Barnes JL, Schilling BK, Falvo MJ, Weiss LW, Creasy AK, Fry AC. Relationship of jumping and agility performance in female volleyball athletes. J Strength Cond Res. 2007 Nov;21(4):1192-6. doi: 10.1519/R-22416.1. PMID 18076276
- [Background] Garcia-de-Alcaraz A, Ramirez-Campillo R, Rivera-Rodriguez M, Romero-Moraleda B. Analysis of jump load during a volleyball season in terms of player role. J Sci Med Sport. 2020 Oct;23(10):973-978. doi: 10.1016/j.jsams.2020.03.002. Epub 2020 Mar 12. PMID 32303475
- [Background] Sheppard JM, Gabbett TJ, Stanganelli LC. An analysis of playing positions in elite men's volleyball: considerations for competition demands and physiologic characteristics. J Strength Cond Res. 2009 Sep;23(6):1858-66. doi: 10.1519/JSC.0b013e3181b45c6a. PMID 19675472